CLINICAL TRIAL: NCT03747861
Title: An Open Clinical Study of Measuring Accuracy of RR- Intervals and Determining the Heart Rate Variability With a Wristband for Registration of ECG RR Intervals for One Hand, SenceBand Compared to the Holter Monitor.
Brief Title: Measuring Accuracy of Wristband for Registration of ECG RR-Intervals for One Hand, SenceBand in Comparison to Holter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Planexta, Inc (Industry)
Collaborators: Pharmaxi LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SenceBand-001
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: HRV
Keywords: R-R intervals; Heart rate; HRV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm for HRV monitoring (Other): For monitoring HRV each subject will put Wristband for registration of ECG RR intervals for one hand, SenceBand in the left wrist and Holter monitor electrodes will be placed in standard configurations places.
  Interventions: Device: SenceBand

INTERVENTIONS:
Device: SenceBand — Wristband for registration of ECG RR intervals for one hand, SenceBand will collect data from 5-minutes intervals each 30 minute within 24 hours

SUMMARY:
The purpose of the study is to evaluate the measuring accuracy of the Wristband for registration of ECG RR intervals for one hand, SenceBand icompared to the Holter monitor (LabTech Ltd).

DETAILED DESCRIPTION:
Non-randomized, prospective, open clinical trial . The main purpose is to evaluate the measuring accuracy of the Wristband for registration of ECG RR intervals for one hand, SenceBand in real-world condition during 24-hours of routine duties in comparison to a predicate device (Holter monitor). For monitoring HRV each subject will put heart rate monitor SenceBand in the randomly assigned wrist and Holter monitor electrodes will be placed in standard configurations places. Data will be collected during routine duties. SenceBand will collect data from 5-minutes intervals each 30 minutes, Holter will collect data continuously over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent;
2. Subject is male or female, aged 18-75;
3. Subject has understood and complied with the requirements of the study protocol and;
4. Subject is fluent in Ukrainian.

Exclusion Criteria:

1. Subject has cardiac pacemakers;
2. Subject is a pregnant woman;
3. Subject has an allergy on polyurethane;
4. Subject refers to vulnerable groups of the population;
5. In investigator's opinion subject is not able physically or intellectually to fulfill the requirements of protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
RR interval accuracy | 5-minute intervals every 30 minutes within 24 hours
  Accuracy of RR intervals estimating

SECONDARY OUTCOMES:
RR-intervals passing | 5-minute intervals every 30 minutes within 24 hours of use
  Frequency of passing of determination of RR-intervals
HRV accuracy for time-domain measures | 5-minute intervals every 30 minutes within 24 hours
  HRV accuracy for time-domain measures (MeanNN, SDNN, RMSSD, pNN50)
HRV accuracy for frequency-domain measures | 5-minute intervals every 30 minutes within 24 hours
  HRV accuracy for time-domain measures (VLF, LF, HF, LF / HF)
HRV accuracy for time-domain measures | 24 hours intervals
  HRV accuracy for time-domain measures (MeanNN, SDNN, RMSSD, pNN50)
HRV accuracy for frequency-domain measures | 24 hours intervals
  HRV accuracy for time-domain measures (VLF, LF, HF, LF / HF)

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Kuznetsova-Arabuli, MD, Principal Investigator — Dr. Sam LLC
Locations (1):
- Doctor Sam Medical Network, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: No